CLINICAL TRIAL: NCT06929208
Title: Investigating the Association Between Heart Rate Variability and Music Listening Prior to Procedures: A Pilot Cohort Study
Brief Title: Heart Rate Variability and Music Listening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/2930a
Record Dates: First submitted 2024-11-05; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Heart Rate Variability; Anxiety; Depression
Keywords: Anxiety; Depression; Heart rate variability
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Electrocardiography; Monitoring, Physiologic

STUDY DESIGN:
Intervention Model Description: Music listening and HRV measurements
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm for HRV and music listening (Experimental): ECG recording for HRV data before, during and after music listening
  Interventions: Device: Electrocardiogram (ECG) monitor; Other: Music listening

INTERVENTIONS:
Device: Electrocardiogram (ECG) monitor — A novel AI-based risk stratification algorithm incorporated into portable platform will be used to monitor and measure patient's ECG, blood pressure, SpO2, and HRV parameters. The platform comprises a tablet application that the clinicians interface with, and coupled with a patient monitoring device with the app that received the real-time patient vital signs to be processed. It requires only a 5-minute 12-lead ECG recording and provides a diagnostic report and risk score on major adverse cardiac events in patients with chest pain complaints. The device is approved as a Class C Medical device by Health Science Authority Singapore for clinical use in Singapore.
  Three ECG samples for HRV data will be recorded before, during and after music listening, with a sampling rate of 1000Hz, 5-10-minute duration in the supine position and breathing spontaneously to minimise influence from external factors.
Other: Music listening — Patients will be given a mobile phone to choose their preferred music to be played during surgery. The music list contains songs across pre-saved playlists spanning different music genres compiled by the institution's music therapist to ensure adequate coverage of the various music genres and to promote relaxation and serenity.

SUMMARY:
High anxiety levels may lead to negative outcomes, and previous studies have shown that music listening could reduce periprocedural anxiety and depression. Recent evidence suggests that a lower heart rate variability (HRV) may be associated with anxiety and depression disorders, but the association of these HRV parameters with preoperative mood in the procedural settings are less defined.

In this prospective cohort pilot study, the study team will investigate the association between HRV and psychological vulnerability (anxiety, depression) in the presence of music listening before procedures. A total of 120 patients about to undergo procedures (surgery, procedures) will be recruited in three healthcare institutions in Singapore (KK Women's and Children's Hospital, Singapore General Hospital, Changi General Hospital). Patients will be asked to have their ECG readings recorded before, during, and after music listening. Preprocedural information (e.g., demographic, clinical) and psychological scores will be collected.

DETAILED DESCRIPTION:
Autonomic nervous system (ANS) comprises two opposing components: sympathetic nervous system (SNS) and parasympathetic nervous system (PNS). It is reported that alterations in the balance between SNS and PNS activity may be related to anxiety and depression. SNS and PNS activity can be non-invasively quantified using HRV, the fluctuation in time intervals between adjacent heartbeats. HRV may be obtained from ECG readings to derive the indices of the variability in time and frequency domains. A meta-analysis in patients with anxiety disorders demonstrated that HRV parameters including root mean square of successive differences (rMSSD), standard deviation, and high frequency HRV (HF-HRV, 0.15-0.4Hz) was lower as compared with healthy individuals.

Compared to the conventional use of pharmacological drugs, music listening is proven to be safer and more cost-effective, reduce perioperative pain, and improve patient satisfaction. Furthermore, music listening can modulate the patient's inflammatory response to reduce anxiety, which could help distracting patients from focusing on negative thoughts of the impending surgery, a major source of anxiety. By providing a source of serenity and calmness through music, patients can divert their attention to and focus less on feelings of anxiety and fear.

The study team therefore proposes to record HRV parameters before, during and after music listening and compare the readings against the psychological scores collected as part of the study. This would facilitate the understanding in the association between HRV and psychological aspects in surgical settings. The overall aim is to develop an individualised, targeted approach to understand the relationship between HRV and mood, and how the improvement in HRV parameters in the presence of music listening may help to improve perioperative experiences.

ELIGIBILITY:
Inclusion Criteria:

1. America Society of Anaesthesiologist (ASA) 1 to 3 adults undergoing procedures (surgery, pain procedures);
2. Able to read and understand English and/or Chinese;
3. Not receiving opioid prior to the procedures.

Exclusion Criteria:

1. With chronic pain;
2. Opioid and drug abuse;
3. Scheduled postoperative Intensive care unit (ICU) admission;
4. With baseline non-sinus heart rhythm or on pacemaker support.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative Heart rate variability (HRV) before, during and after music listening - root mean square of successive differences NN intervals (rMSSD) | 1 day
  Preoperative HRV parameters on root mean square of successive differences NN intervals (rMSSD) will be collected before, during and after music listening, with a sampling rate of 1000Hz, 5-10-minutes duration.
Preoperative Heart rate variability (HRV) before, during and after music listening - low frequency (LF)-HRV | 1 day
  Preoperative HRV parameters on low frequency (LF)-HRV will be collected before, during and after music listening, with a sampling rate of 1000Hz, 5-10-minutes duration.
Preoperative Heart rate variability (HRV) before, during and after music listening - High Frequency (HF)-HRV | 1 day
  Preoperative HRV parameters on High Frequency (HF)-HRV will be collected before, during and after music listening, with a sampling rate of 1000Hz, 5-10-minutes duration.
Preoperative Heart rate variability (HRV) before, during and after music listening - LF/HF ratio | 1 day
  Preoperative HRV parameters on LF/HF ratio will be collected before, during and after music listening, with a sampling rate of 1000Hz, 5-10-minutes duration.

SECONDARY OUTCOMES:
Preoperative anxiety before and after music listening | 1 day
  Before and after music listening, a visual analogue scale depicting anxiety (VAS-A) comprises a 10 cm line will be administered, on which the participant marks the current degree of anxiety with the left end of the line being labelled "no anxiety" and the right end being labelled "maximum anxiety".
Preoperative depression score before and after music listening | 1 day
  Before and after music listening, depression score will also be collected via Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 consists of 9 questions about the patient's feelings, with each question scored from 0 to 3 based on the frequency of symptom; hence having a total score ranging from 0 to 27. Scores of 0 to 4 depicts no depression, whereas 5 to 9 may indicate a mild depression. 10 and above will indicate moderate/severe depression.

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - Changi General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
To be shared upon request